CLINICAL TRIAL: NCT01260142
Title: A Randomized, Open-Label, Single-Bolus, 2-Period, Multi-Dose Level, 3 Cohort Crossover Design, Pharmacokinetic/Pharmacodynamic Study of Lusedra (Fospropofol Disodium) Injection Compared With Propofol Injectable Emulsion
Brief Title: A PK/PD Study of Fospropofol Disodium Compared With Propofol Injectable Emulsion
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: E2083-A001-410
Record Dates: First submitted 2010-12-13; First posted 2010-12-15 (Estimated); Results first posted 2017-01-27 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2016-11

CONDITIONS: Anesthesia
MeSH Terms: interventions — fospropofol; Propofol

ARMS (3):
- Arm 1 (Experimental)
  Interventions: Drug: Fospropofol disodium, propofol
- Arm 2 (Experimental)
  Interventions: Drug: Fospropofol disodium, propofol
- Arm 3 (Experimental)
  Interventions: Drug: Fospropofol disodium, propofol

INTERVENTIONS:
Drug: Fospropofol disodium, propofol — Two Treatment Periods: fospropofol disodium 6.5 mg/kg single intravenous (IV) bolus followed by propofol injectable emulsion 0.65 mg/kg IV bolus, or propofol injectable emulsion 0.65 mg/kg IV bolus followed by fospropofol disodium 6.5 mg/kg IV bolus.
  Arms: Arm 1
Drug: Fospropofol disodium, propofol — Two Treatment Periods: fospropofol disodium 10.0 mg/kg single intravenous (IV) bolus followed by propofol injectable emulsion 1.0 mg/kg IV bolus, or propofol injectable emulsion 1.0 mg/kg IV bolus followed by fospropofol disodium 10.0 mg/kg IV bolus.
  Arms: Arm 2
Drug: Fospropofol disodium, propofol — Two Treatment Periods: fospropofol disodium 15.0 mg/kg single intravenous (IV) bolus followed by propofol injectable emulsion 1.5 mg/kg IV bolus, or propofol injectable emulsion 1.5 mg/kg IV bolus followed by fospropofol disodium 15.0 mg/kg IV bolus.
  Arms: Arm 3

SUMMARY:
This study is designed to characterize the pharmacokinetic and pharmacodynamic effect of fospropofol disodium in comparison to propofol. In addition, the study will compare the maximum sedative effect, safety and tolerability of fospropofol disodium and propofol.

ELIGIBILITY:
Inclusion

* Males or females greater than or equal to 18 or less than or equal to 45 years old
* Non-smokers for at least 18 months prior to Screening
* Body Mass Index (BMI) less than or equal to 30 Exclusion
* Subjects having a past or current medical history of any respiratory illness including asthma
* Subjects currently taking any medications (birth control will be allowed if the subject has been taking it for at least 12 weeks prior to dosing and during the entire study), including over-the-counter (OTC) medication, within 14 days of Screening
* Subjects with a known or suspected history of drug or alcohol misuse within 6 months prior to Screening, or who have a positive urine drug test at Screening and pre-dose at Visit 2 and Visit 3
* Subjectw who are allergic to eggs, egg products, soybeans, or soy products
* Subjects with a positive pregnancy test at Screening or breastfeeding
* Subjects who are unwilling or unable to abide by the requirements of the study
* Subjects who have any condition that would make him/her, in the opinion of the investigator, unsuitable for the study or who, in the opinion of the investigator, are not likely to complete the study for any reason

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2010-11; Primary Completion 2011-02 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Randi Fain, Study Director — Eisai Inc.
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Each cohort had 2 treatment periods that were separated by a 7 to 14 day washout: fospropofol disodium, followed by propofol injectable emulsion; or propofol injectable emulsion, followed by fospropofol disodium.
Groups:
- Cohort 1 (Sequence A): Participants were administered intravenous (IV) bolus of 6.5 mg/kg of fospropofol disodium during Treatment Period 1, then after a 7-14 day washout began Treatment Period 2 with an IV bolus of 0.65 mg/kg propofol injectable emulsion.
- Cohort 1 (Sequence B): Participants were administered an IV bolus of 0.65 mg/kg of propofol injectable emulsion during Treatment Period 1, then after a 7-14 day washout began Treatment Period 2 with an IV bolus of 6.5 mg/kg of fospropofol disodium.
- Cohort 2 (Sequence C): Participants were administered an IV bolus of 10 mg/kg of fospropofol disodium during Treatment Period 1, then after a 7-14 day washout began Treatment Period 2 with an IV bolus of 1.0 mg/kg propofol injectable emulsion.
- Cohort 2 (Sequence D): Participants were administered an IV bolus of 1.0 mg/kg of propofol injectable emulsion during Treatment Period 1, then after a 7-14 day washout began Treatment Period 2 with an IV bolus of 10 mg/kg of fospropofol disodium.
- Cohort 3 (Sequence E): Participants were administered an IV bolus of 15 mg/kg of fospropofol disodium during Treatment Period 1, then after a 7-14 day washout began Treatment Period 2 with an IV bolus of 1.5 mg/kg propofol injectable emulsion.
- Cohort 3 (Sequence F): Participants were administered an intravenous IV bolus of 1.5 mg/kg of propofol injectable emulsion during Treatment Period 1, then after a 7-14 day washout began Treatment Period 2 with an IV bolus of 15 mg/kg of fospropofol disodium.
Period: Treatment Period 1
Arm/Group | Cohort 1 (Sequence A) | Cohort 1 (Sequence B) | Cohort 2 (Sequence C) | Cohort 2 (Sequence D) | Cohort 3 (Sequence E) | Cohort 3 (Sequence F)
Started | 6 | 6 | 6 | 6 | 6 | 6
Completed | 5 | 5 | 6 | 6 | 4 | 3
Not Completed | 1 | 1 | 0 | 0 | 2 | 3
Not completed — Study on hold | 1 | 1 | 0 | 0 | 1 | 2
Not completed — Unexplained elevated sys. BP | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1
Period: Treatment Period 2
Arm/Group | Cohort 1 (Sequence A) | Cohort 1 (Sequence B) | Cohort 2 (Sequence C) | Cohort 2 (Sequence D) | Cohort 3 (Sequence E) | Cohort 3 (Sequence F)
Started | 5 | 5 | 6 | 6 | 4 | 3
Completed | 5 | 5 | 6 | 6 | 4 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cohort 1 (Sequence A): Participants were administered an intravenous (IV) bolus of 6.5 mg/kg of fospropofol disodium during Treatment Period 1, then after a 7-14 day washout began Treatment Period 2 with an IV bolus of 0.65 mg/kg propofol injectable emulsion.
- Cohort 3 ( Sequence F): Participants were administered an IV bolus of 1.5 mg/kg of propofol injectable emulsion during Treatment Period 1, then after a 7-14 day washout began Treatment Period 2 with an IV bolus of 15 mg/kg of fospropofol disodium.
- Total: Total of all reporting groups
Arm/Group | Cohort 1 (Sequence A) | Cohort 1 (Sequence B) | Cohort 2 (Sequence C) | Cohort 2 (Sequence D) | Cohort 3 (Sequence E) | Cohort 3 ( Sequence F) | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 36
Age, Continuous [Mean (Standard Deviation); unit: Years] | 22.3 (1.51) | 25.5 (3.78) | 25.3 (4.46) | 22.7 (2.88) | 29 (4.34) | 23.8 (3.37) | 24.8 (3.98)
Gender [Count of Participants; unit: Participants]
  Female | 2 | 2 | 3 | 2 | 2 | 4 | 15
  Male | 4 | 4 | 3 | 4 | 4 | 2 | 21

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Time 0 to Infinity of Fospropofol (AUC(0-inf))
Description: AUC(0-inf) is a measure of drug concentration equal to the area under the plasma concentration-time profile from time 0 to infinity. An arterial line (A-line) and venous line (V-line) were placed prior to dosing during each treatment period and used to collect blood samples for plasma concentration measurements at specific time points. Plasma arterial and venous concentrations of fospropofol were quantified by high-performance liquid chromatography with mass spectrometric detection (LC-MS/MS). The AUC(0-inf) was calculated from the sum of AUC from time 0 to time t (AUC(0-t)) and the residual area calculated as Ct/λz, where Ct was the observed concentration at last quantifiable concentration and λz was the terminal elimination rate constant. The plasma concentrations from the venous sampling were descriptively compared head-to-head with the arterial sampling.
Time Frame: Days 1, and 7-14 (Arterial Sample: Pre-dose, and 0.5, 1, 1.5, 2, 4, 8, 16, 30, 45, 60, 120, 180, 240, 300, and 360 minutes post-dose. Venous Sample: Pre-dose, and 1, 4, and 30 minutes post-dose).
Population: Pharmacokinetic (PK) Analysis Set is the group of participants who have sufficient pharmacokinetic data to derive at least one PK parameter.
Measure: Mean (Standard Deviation); unit: ug.h/L
Groups:
- Fospropofol 6.5 mg/kg: Cohort 1: participants were administered an intravenous (IV) bolus of 6.5 mg/kg of fospropofol disodium during Treatment Period 1 (Sequence Group A) or Treatment Period 2 (Sequence Group B).
- Fospropofol 10 mg/kg: Cohort 2: participants were administered an IV bolus of 10 mg/kg of fospropofol disodium during Treatment Period 1 (Sequence Group C) or Treatment Period 2 (Sequence Group D).
- Fospropofol 15 mg/kg: Cohort 3: participants were administered an IV bolus of 15 mg/kg of fospropofol disodium during Treatment Period 1 (Sequence Group E) or Treatment Period 2 (Sequence Group F).
Arm/Group | Fospropofol 6.5 mg/kg | Fospropofol 10 mg/kg | Fospropofol 15 mg/kg
Number analyzed (Participants) | 10 | 10 | 7
ug.h/L | 16522 (3639.1) | 25052 (5923.8) | 36629 (5903.3)

2. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Time 0 to Infinity of Propofol
Description: An A-line and V-line were placed prior to dosing during each treatment period and used to collect blood samples for plasma concentration measurements at specific time points. Plasma arterial and venous concentrations of propofol were quantified by high-performance liquid chromatography with mass spectrometric detection (LC-MS/MS). The AUC(0-inf) was calculated from the sum of AUC(0-t) and the residual area calculated as Ct/λz, where Ct was the observed concentration at last quantifiable concentration and λz was the terminal elimination rate constant. The plasma concentrations from the venous sampling were descriptively compared head-to-head with the arterial sampling. In addition, the arterial plasma concentrations of fospropofol, propofol liberated from fospropofol, and propofol delivered from propofol injectable emulsion were used to refine the population PK model developed previously.
Time Frame: as for outcome 1
Population: PK Analysis Set
Measure: Mean (Standard Deviation); unit: ug.h/L
Groups:
- Fospropofol 6.5 mg/kg: Cohort 1: participants were administered an IV bolus of 6.5 mg/kg of fospropofol disodium during Treatment Period 1 (Sequence Group A) or Treatment Period 2 (Sequence Group B).
- Propofol 0.65 mg/kg: Cohort 1: participants were administered an IV bolus of 0.65 mg/kg of propofol injectable emulsion during Treatment Period 1 (Sequence Group B) or Treatment Period 2 (Sequence Group A).
- Propofol 1.0 mg/kg: Cohort 2: participants were administered an IV bolus of 1.0 mg/kg of propofol injectable emulsion during Treatment Period 1 (Sequence Group D) or Treatment Period 2 (Sequence Group C).
- Propofol 1.5 mg/kg: Cohort 3: participants were administered an IV bolus of 1.5 mg/kg of propofol injectable emulsion during Treatment Period 1 (Sequence Group F) or Treatment Period 2 (Sequence Group E).
Arm/Group | Fospropofol 6.5 mg/kg | Propofol 0.65 mg/kg | Fospropofol 10 mg/kg | Propofol 1.0 mg/kg | Fospropofol 15 mg/kg | Propofol 1.5 mg/kg
Number analyzed (Participants) | 9 | 5 | 7 | 5 | 4 | 4
ug.h/L | 1541 (224.7) | 467 (88.3) | 2368 (435.3) | 661 (147.3) | 3807 (466.2) | 893 (127.7)

3. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Time 0 to Time t (AUC(0-t)) of Fospropofol
Description: Arterial and venous blood samples were collected and analyzed for fospropofol concentrations as described previously. AUC(0-t) was calculated using the log-linear trapezoidal rule (linear trapezoidal rule up to maximum observed plasma concentration (Cmax), log trapezoidal rule following Cmax) from time of dosing to the last quantifiable concentration. The plasma concentrations from the venous sampling were descriptively compared head-to-head with the arterial sampling.
Time Frame: as for outcome 1
Population: PK Analysis Set
Measure: Mean (Standard Deviation); unit: ug.h/L
Arm/Group | Fospropofol 6.5 mg/kg | Fospropofol 10 mg/kg | Fospropofol 15 mg/kg
Number analyzed (Participants) | 10 | 10 | 8
ug.h/L | 16046 (3439.6) | 24473 (5729.5) | 36330 (5488.7)

4. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Time 0 to Time t of Propofol
Description: Arterial and venous blood samples were collected and analyzed for propofol concentrations as described previously. AUC(0-t) was calculated using the log-linear trapezoidal rule (linear trapezoidal rule up to Cmax, log trapezoidal rule following Cmax) from time of dosing to the last quantifiable concentration. The plasma concentrations from the venous sampling were descriptively compared head-to-head with the arterial sampling. In addition, the arterial plasma concentrations of fospropofol, propofol liberated from fospropofol, and propofol delivered from propofol injectable emulsion were used to refine the population PK model developed previously.
Time Frame: as for outcome 1
Population: PK Analysis Set
Measure: Mean (Standard Deviation); unit: ug.h/L
Arm/Group | Fospropofol 6.5 mg/kg | Propofol 0.65 mg/kg | Fospropofol 10 mg/kg | Propofol 1.0 mg/kg | Fospropofol 15 mg/kg | Propofol 1.5 mg/kg
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 8 | 8
ug.h/L | 1343 (166.9) | 385 (84.5) | 2009 (413.9) | 578 (107.2) | 3019 (468.2) | 801 (141.6)

5. Primary Outcome: Maximum Drug Plasma Concentration (Cmax) of Fospropofol
Description: Arterial and venous blood samples were collected and analyzed for fospropofol concentrations as described previously. Cmax was the highest plasma drug concentration observed over the entire sampling period, and was obtained directly from the experimental plasma concentration time data without interpolation. The plasma concentrations from the venous sampling were descriptively compared head-to-head with the arterial sampling.
Time Frame: as for outcome 1
Population: PK Analysis Set
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Fospropofol 6.5 mg/kg | Fospropofol 10 mg/kg | Fospropofol 15 mg/kg
Number analyzed (Participants) | 10 | 10 | 8
ug/mL | 95.6 (16.45) | 146.3 (25.6) | 207.3 (29.17)

6. Primary Outcome: Maximum Drug Plasma Concentration of Propofol
Description: Arterial and venous blood samples were collected and analyzed for propofol concentrations as described previously. Cmax was the highest plasma drug concentration observed over the entire sampling period, and was obtained directly from the experimental plasma concentration time data without interpolation. The plasma concentrations from the venous sampling were descriptively compared head-to-head with the arterial sampling.
Time Frame: as for outcome 1
Population: PK Analysis Set
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Fospropofol 6.5 mg/kg | Propofol 0.65 mg/kg | Fospropofol 10 mg/kg | Propofol 1.0 mg/kg | Fospropofol 15 mg/kg | Propofol 1.5 mg/kg
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 8 | 8
ug/mL | 1.5 (0.47) | 8 (6) | 2.1 (0.74) | 8.6 (6.39) | 3.1 (0.7) | 9.5 (4.44)

7. Secondary Outcome: Maximal Sedative Effect Using the Bispectral Index (BIS) Score
Description: Pharmacodynamic (PD) effects were obtained from continuous BIS score recordings obtained throughout the study and from clinical assessment of sedation using the Modified Observer's Assessment of Alertness/Sedation (MOAA/S) scale. The BIS measurements continued until the participant was fully recovered in the opinion of the investigator or until the PD effect measure returned to baseline. The BIS score varied between 100 (associated with being fully awake) and 0 (associated with a flat line on the electroencephalogram (EEG)). The BIS Index was described by the maximal effect (Emax) model.
Time Frame: Days 1, and 7-14 (BIS measurements were to continue until the subject was fully recovered in the opinion of the investigator or until the PD effect measures returned to baseline measures)
Population: PD analysis set included all participants who had sufficient PD data to derive at least one PD assessment.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Fospropofol 6.5 mg/kg | Propofol 0.65 mg/kg | Fospropofol 10 mg/kg | Propofol 1.0 mg/kg | Fospropofol 15 mg/kg | Propofol 1.5 mg/kg
Number analyzed (Participants) | 11 | 11 | 12 | 12 | 9 | 10
Scores on a scale | 70.2 (10.3) | 81.5 (8.12) | 55.4 (11.35) | 65.8 (15.17) | 38.6 (7.78) | 49 (10.1)

8. Secondary Outcome: Maximal Sedative Effect Using the Modified Observer's Assessment of Alertness/Sedation Scale
Description: PD effects were determined from continuous BIS score recordings and from clinical assessment of sedation using the MOAA/S scale. The MOAA/S scale was used to rate the level of alertness/sedation from a score of 0 (does not respond to painful stimulus) to 5 (alert) in the category of responsiveness, with 5 being the MOAA/S value for a fully awake adult. Time to sedation was defined as the time from the first dose of study medication to the first two consecutive MOAA/S scores less than or equal to 4. Fully awake status was reached at the first of 3 consecutive MOAA/S scores of 5 measured every 2 minutes after study drug administration. The MOAA/S scale was described by the Emax model.
Time Frame: Days 1, and 7-14 (2 minutes prior to study drug administration and every 2 minutes thereafter for 20 minutes or until the subject reached Fully Alert status, whichever was later).
Population: PD Analysis Set
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Fospropofol 6.5 mg/kg | Propofol 0.65 mg/kg | Fospropofol 10 mg/kg | Propofol 1.0 mg/kg | Fospropofol 15 mg/kg | Propofol 1.5 mg/kg
Number analyzed (Participants) | 11 | 11 | 12 | 12 | 9 | 10
Scores on a scale | 4.1 (1.58) | 4.7 (0.65) | 2.8 (1.64) | 3.9 (1.44) | 0.3 (0.71) | 1.7 (1.57)

9. Secondary Outcome: Relative Bioavailability of Fospropofol and Propofol
Description: The PK parameters for propofol from propofol injectable emulsion were used as the reference formulation. Because propofol is a metabolite of fospropofol, all calculations were conducted after correcting for the different molecular weights of these formulations. Molecular weights of 332.24 (288.24 for free base) and 178.27 were used for fospropofol disodium and propofol injectable emulsion, respectively. The propofol parameters were adjusted as appropriate as discussed above and natural log transformed prior to comparison. Relative bioavailability of propofol from fospropofol disodium (E2083) to propofol from propofol injectable emulsion is calculated as (AUC(FP) x Total Dose of Propofol/AUC(P) x Total Dose of E2083) x Molecular fraction, where AUC(FP) is AUC(0-t) or AUC(0-inf) of propofol from E2083, AUC(P) is AUC(0-t) or AUC(0-inf) of propofol from propofol injectable emulsion and molecular fraction is molecular weight of propofol (178.27)/E2083 (332.24).
Time Frame: as for outcome 1
Population: PK Analysis Set
Measure: Mean (Standard Deviation); unit: ng x hr/mL
Groups:
- Cohort 1 (Fospropofol 6.5 : Propofol 0.65): Cohort 1 (Sequence A): participants were administered an IV bolus of 6.5 mg/kg of fospropofol disodium during Treatment Period 1, then after a 7-14 day washout began Treatment Period 2 with an IV bolus of 0.65 mg/kg propofol injectable emulsion.
  Cohort 1: Sequence B: participants were administered an IV bolus of 0.65 mg/kg of propofol injectable emulsion during Treatment Period 1, then after a 7-14 day washout began Treatment Period 2 with an IV bolus of 6.5 mg/kg of fospropofol disodium.
- Cohort 2 (Fospropofol 10.0 : Propofol 1.0): Cohort 2 (Sequence C): Participants were administered an IV bolus of 10 mg/kg of fospropofol disodium during Treatment Period 1, then after a 7-14 day washout began Treatment Period 2 with an IV bolus of 1.0 mg/kg propofol injectable emulsion.
  Cohort 2 (Sequence D): Participants were administered an IV bolus of 1.0 mg/kg of propofol injectable emulsion during Treatment Period 1, then after a 7-14 day washout began Treatment Period 2 with an IV bolus of 10 mg/kg of fospropofol disodium.
- Cohort 3 (Fospropofol 15.0 : Propofol 1.5): Cohort 3 (Sequence E): participants were administered an IV bolus of 15 mg/kg of fospropofol disodium during Treatment Period 1, then after a 7-14 day washout began Treatment Period 2 with an IV bolus of 1.5 mg/kg propofol injectable emulsion.
  Cohort (Sequence F): participants were administered an IV bolus of 1.5 mg/kg of propofol injectable emulsion during Treatment Period 1, then after a 7-14 day washout began Treatment Period 2 with an IV bolus of 15 mg/kg of fospropofol disodium.
Arm/Group | Cohort 1 (Fospropofol 6.5 : Propofol 0.65) | Cohort 2 (Fospropofol 10.0 : Propofol 1.0) | Cohort 3 (Fospropofol 15.0 : Propofol 1.5)
Number analyzed (Participants) | 10 | 10 | 7
ng x hr/mL
  AUC(0-t) | 0.684 (0.1505) | 0.661 (0.0987) | 0.713 (0.0671)
  AUC(0-inf) | 0.694 (0.0882) | 0.68 (0.0495) | 0.836 (0.0198)

ADVERSE EVENTS:
Time Frame: An adverse event in Treatment Period 1 was counted up to 3 days after the first treatment; an adverse event in Treatment Period 2 was counted up to 3 days after the second treatment. Up to approximately 32 days.
Description: A subject with 2 or more adverse events in the same System Organ Class was counted only once for that System Organ Class (or Preferred Term).
Arm/Group | Fospropofol 6.5 mg/kg | Propofol 0.65 mg/kg | Fospropofol 10 mg/kg | Propofol 1.0 mg/kg | Fospropofol 15 mg/kg | Propofol 1.5 mg/kg
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11 | 0/12 | 0/12 | 0/9 | 0/10
Other Adverse Events (participants affected / at risk) | 8/11 | 5/11 | 9/12 | 4/12 | 6/9 | 2/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fospropofol 6.5 mg/kg (N=11) | Propofol 0.65 mg/kg (N=11) | Fospropofol 10 mg/kg (N=12) | Propofol 1.0 mg/kg (N=12) | Fospropofol 15 mg/kg (N=9) | Propofol 1.5 mg/kg (N=10)
Feeling hot (General disorders) | 0 | 0 | 1 | 1 | 0 | 0
Burning sensation (Nervous system disorders) | 2 | 1 | 0 | 1 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 1 | 1 | 0 | 0
Mental impairment (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 3 | 1 | 3 | 0
Genital burning sensation (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 1 | 0
Pruritus genital (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 1 | 0
Apnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2 | 0 | 1 | 2
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 3 | 3 | 0 | 1 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 3 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other